CLINICAL TRIAL: NCT04284904
Title: Role of aGVHD Biomarkers on aGVHD Risks in Patients Underwent Hematopoietic Stem Cell Transplantation
Brief Title: Role of aGVHD Biomarkers on aGVHD Risks
Acronym: GVHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Other Study IDs: S2019-177-02
Record Dates: First submitted 2020-01-30; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: GVHD,Acute; Biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- matched sibling hematopoietic stem cell transplantation: aGVHD biomarker in matched sibling donor hematopoietic stem cell transplantation
  Interventions: Diagnostic Test: aGVHD biomarker
- unrelated allogeneic hematopoietic stem cell transplantation: aGVHD biomarker in unrelated donor hematopoietic stem cell transplantation
  Interventions: Diagnostic Test: aGVHD biomarker
- haploidentical hematopoietic stem cell transplantation: aGVHD biomarker in haploidentical donor hematopoietic stem cell transplantation
  Interventions: Diagnostic Test: aGVHD biomarker

INTERVENTIONS:
Diagnostic Test: aGVHD biomarker — To verify the effectiveness of aGVHD biomarkers monitoring in predicting aGVHD risks

SUMMARY:
To establish risk rating criteria of biological protein marker, determine the role and consistency of aGVHD biomarkers in aGVHD diagnosis and aGVHD prognosis, and evaluate the the impact on non-relapse mortality and relapse and disease free survival, the multicenter study on aGVHD biomarkers detection in the patients underwent allogeneic hematopoietic stem cell transplantation was performed.

DETAILED DESCRIPTION:
1. To establish standard risk rating criteria of aGVHD biomarkers;
2. To verify the role of aGVHD biomarkers monitored in predicting aGVHD risks;
3. To determine the correlation between aGVHD biomarkers monitored and aGVHD risk;
4. To carry out a observative study in patients with aGVHD treatment about therapeutic protocols and medication efficacy;
5. To predict the correlation between the high-risk patients with aGVHD and non-relapse mortality and disease free survival;

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hematological diseases.
2. Have underwent first allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies.

Exclusion Criteria:

1. recipients of second allogeneic stem cell transplant.
2. pregnant or breast-feeding women.
3. Serum creatinine > 2.0 mg/dL or creatinine clearance < 40 mL/min measured or calculated by Cockroft-Gault equation.
4. human immunodeficiency virus infection
5. active hepatitis b virus, hepatitis C virus infection and need antivirus treatment.
6. Subjects with evidence of relapsed primary disease, or subjects who have been treated for relapse after the allo-HSCT was performed, or graft rejection.
7. allergic history to Janus kinase inhibitors.
8. Severe organ dysfunction unrelated
9. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.

Max Age: 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosed with hematological diseases and nderwent first allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The correlation between cumulative incidence of aGVHD relapse at 3 months after transplantation with aGVHD biomarkers monitored (serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 14 days after stem cell infusion
  For all cytokines/biomarkers (serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R)) that are measured by flow cytometry repeatedly over time(every two week until three months after transplantation), a nonparametric smoothing plot will be produced in the first step to view changes in the trend. Expression level changes on the onset of aGVHD from baseline measures will be correlated with aGVHD relapse at 3 months after transplantation.

SECONDARY OUTCOMES:
The correlation between cumulative incidence of cGVHD relapse at 24 months after transplantation with aGVHD biomarkers monitored(serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 14 days after stem cell infusion
  For all cytokines/biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) that are measured repeatedly over time (every two week until three months after transplantation), a nonparametric smoothing plot will be produced in the first step to view changes in the trend. Expression level changes on the onset of aGVHD from baseline measures will be correlated with cGVHD relapse at 24 months after transplantation
The correlation between cumulative incidence of relapsed aGVHD grade at 3 months after transplantation with aGVHD biomarkers monitored(serum concentration of REG3a; ST22; IL-6; IL-8;TNF R1 | 14 days after stem cell infusion
  For all cytokines/biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) that are measured repeatedly over time (every two week until three months after transplantation), a nonparametric smoothing plot will be produced in the first step to view changes in the trend. Expression level changes on the onset of aGVHD from baseline measures will be correlated with relapsed aGVHD grade (1, 2, 3, 4) at 3 months after transplantation
The correlation between overall survival with aGVHD biomarkers monitored(serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 14 days after stem cell infusion
  Expression level changes of aGVHD biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) on the onset of aGVHD from baseline measures will be correlated with overall survival
The correlation between relapse free survival with aGVHD biomarkers monitored(serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 14 days after stem cell infusion
  Expression level changes of aGVHD biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) on the onset of aGVHD from baseline measures will be correlated with relapse free survival
The correlation between non relapse mortality with aGVHD biomarkers monitored(serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 14 days after stem cell infusion
  Expression level changes of aGVHD biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) on the onset of aGVHD from baseline measures will be correlated with non relapse mortality

OTHER OUTCOMES:
The correlation between cumulative incidence of aGVHD relapse at 3 months after transplantation with aGVHD biomarkers monitored(serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 7 days after aGVHD treatment
  For all cytokines/biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) that are measured repeatedly over time (every two week until three months after transplantation), a nonparametric smoothing plot will be produced in the first step to view changes in the trend. Expression level changes 7 days after aGVHD treatment from baseline measures will be correlated with aGVHD relapse at 3 months after transplantation
The correlation between cumulative incidence of cGVHD relapse at 24 months after transplantation with aGVHD biomarkers monitored(serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 7 days after aGVHD treatment
  For all cytokines/biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) that are measured repeatedly over time (every two week until three months after transplantation), a nonparametric smoothing plot will be produced in the first step to view changes in the trend. Expression level changes 7 days after aGVHD treatment from baseline measures will be correlated with cGVHD relapse at 24 months after transplantation
The correlation between overall survival with aGVHD biomarkers monitored(serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 7 days after aGVHD treatment
  Expression level changes of aGVHD biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) 7 days after aGVHD treatment from baseline measures will be correlated with overall survival
The correlation between non relapse mortality with aGVHD biomarkers monitored(serum concentration of REG3: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) | 7 days after aGVHD treatment
  Expression level changes of aGVHD biomarkers (serum concentration of REG3a: regenerating islet-derived-3-a; ST2: suppression of tumorigenicity 2; IL-6; IL-8; TNF R) 7 days after aGVHD treatment from baseline measures will be correlated with non relapse mortality

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided